CLINICAL TRIAL: NCT03544944
Title: A Prospective, Randomized, Single-blinded (Evaluator), Parallel, Multi-center, Phase 3 Trial in Bowel Preparation for Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taejoon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJP-008-301
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2018-04

CONDITIONS: Bowel Preparation
Keywords: bowel preparation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TJP-008-1 (Experimental)
  Interventions: Drug: TJP-008-1
- TJP-008-2 (Experimental)
  Interventions: Drug: TJP-008-2
- Coolprep powder (Active Comparator)
  Interventions: Drug: Coolprep powder

INTERVENTIONS:
Drug: TJP-008-1 — Subjects who are randomized into group TJP-008-1 will receive bowel preparation on the same-day.
  Arms: TJP-008-1
Drug: TJP-008-2 — Subjects who are randomized into group TJP-008-2 will receive bowel preparation from evening to next morning.
  Arms: TJP-008-2
Drug: Coolprep powder — Subjects who are randomized into group Coolprep will receive bowel preparation from evening to next morning.
  Arms: Coolprep powder

SUMMARY:
This is a prospective randomized study compared with active control arm. The investigators compare the colon cleansing in patients undergoing colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent.
* Male and female outpatients and inpatients aged: ≥19
* Patients BMI shoule be ≤ 30

Exclusion Criteria:

* Patients with past history within last 12 months or current episode of severe constipation
* Known glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Known phenylketonuria.
* Clinically relevant findings on physical examination based on the Investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Ratio of subjects With successful Bowel Cleansing | 1 day of scheduled colonoscopy

SECONDARY OUTCOMES:
Easch segments ratio of subject with successful Bowel Cleansing | 1 day of scheduled colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Taejoon Pharmaceutical Co., Ltd., Seoul, South Korea